CLINICAL TRIAL: NCT04194281
Title: Action Observation Training [AOT] to Improve Upper Limb Function in Infants After Unilateral Brain Lesion - a Feasibility Study
Brief Title: Feasibility of Action Observation Training [AOT] in Infants After Unilateral Brain Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-02028
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Perinatal Brain Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Action Observation Therapy [AOT] (Experimental)
  Interventions: Other: Action Observation Training [AOT]

INTERVENTIONS:
Other: Action Observation Training [AOT] — Parents are instructed to show their child repetitive arm, hand and finger movements in a playful and age-appropriate way for about 20 minutes a day, divided into several short sequences. AOT is to be carried out for four weeks at home by the parents and, if necessary, other caregivers. The parents receive instructions which contain background information on the possible importance of AOT for improving the functions of the upper limb, information about positions, promoting motivation, attention and interest as well as tips for promoting movement observation in everyday life.

SUMMARY:
The study examines whether infants with a perinatal unilateral brain lesion can perform an "Action Observation Training" [AOT] at the age of 9-12 months . AOT is the targeted and concentrated observation of movements and actions to learn new motor skills. In adults with hemiplegia after a stroke and in older children with hemiplegia, AOT can lead to an improvement in the functions of the affected hand/arm. Infants with early unilateral brain damage are at increased risk of developing a hemiplegia and thus impaired upper limb function. There is little known about treatment options to promote arm and hand skills in early childhood and their effectiveness. In particular, there is a lack of knowledge whether AOT could also be used in infants. It is known that even in infants at an early age brain activity can be measured while they are observing movements and infants learn a lot about observing and imitating.

Knowledge about the measurement of manual skills is also reduced. So far, tests have been used to observe and evaluate how infants use their hands when playing (e.g. Mini-Assisting Hand Assessment). The aim of this study is to investigate whether measurements with motion sensors can also be used in infants.

In the pre-post study, about 5 to 10 toddlers will be examined. During four weeks, the parents should give the child 20 minutes of AOT per day at home. A therapy diary will be completed for this purpose. During six weeks, the parents will use movement sensors on two days a week for the upper limb of the infants. Finally, three questionnaires about the AOT and the motion sensors will be completed by the parents.

ELIGIBILITY:
Inclusion Criteria:

* Premature and term-born infants aged 9-12 months
* Perinatal unilateral brain damage due to cerebral hemorrhage or stroke
* Informed consent to study participation by the parents or legal representative

Exclusion Criteria:

* Infants with impaired vision
* Other diagnoses than early childhood brain damage affecting the functions of the upper extremities (e.g. plexus palsy)
* Infants who participate in other studies of upper extremity interventions
* Parents do not understand the study and the intervention due to foreign language skills

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of and adherence to Action Observation Training in infants measured by an intervention diary | Four weeks during the Intervention
  To assess the adherence of the intervention the parents fill out a diary. In addition to the training duration in minutes per day, the number of training sequences, the persons involved, the content of the AOT and the attention, motivation and imitation behaviour of the child should also be documented. The parents are asked to write down further comments on the form which may contribute to a better understanding.

SECONDARY OUTCOMES:
Action Observation Training Questionnaire Part I feasibility | Posttest, expected to be an average of 10 minutes
  The parents fill out a questionnaire about the feasibility of AOT with a minimum score of 0 and a maximum score of 19 (higher score means better feasibility).
Action Observation Training Questionnaire Part II acceptance | Posttest, expected to be an average of 10 minutes
  The parents fill out a questionnaire about their acceptance of AOT with a minimum score of 0 and a maximum score of 24 (higher score means better feasibility).
Hand Assessment for Infants [HAI] | Pre- and Posttest, expected to be an average of 15 minutes
  The HAI ist a descriptive and evaluative assessment of upper limb function for use with infants aged 3 to 12 months at risk of unilateral cerebral palsy. The HAI measures the use of both hands and quantifies a possible asymmetry of hand use. The age-appropriate play situation is recorded on video. The score ranges from 0 to 100 HAI-Units (the higher the score the better the hand function).
Mini-Assisting Hand Assessment [Mini-AHA] | Pre- and Posttest, expected to be an average of 15 minutes
  The Mini-AHA measures and describes how effectively infants with unilateral cerebral palsy at the age of 8 to 18 months use their affected hand in bimanual Play. A semi-structured age-appropriate play situation is recorded on video. The score ranges from 0 to 100 Mini-AHA-Units (the higher the score the better the hand function).
Accelerometry | The infants wear the accelerometers two days a week during the study duration of six weeks
  To measure the quantity of arm movements during the study period, the parents put on movement sensors for each arm of the infant.
Questionnaire Accelerometer | Posttest, expected to be an average of 5 minutes
  To assess the feasibility of accelerometers in infants, the parents fill out a questionnaire about their experience. The score ranges from 0 to 40 (the higher the score the better the result).
System Usability Scale [SUS] | Posttest, expected to be an average of 5 minutes
  To assess the usability of accelerometers, the parents fill out the SUS with questions about their experiences with the system. The scale ranges from 0 to 100 (the higher the score the better the Usability).

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Grunt, PD Dr. med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Kinderklinik Inselspital Bern, Bern, Switzerland